CLINICAL TRIAL: NCT03386539
Title: Phase III Multicenter Open-label Randomized Clinical Trial Comparing Everolimus and Low Dose Tacrolimus to Tacrolimus and Mycophenolate Mofetil at 6 mo Post-Transplant to Prevent Long-term Complications After Pediatric Heart Transplantation
Brief Title: Tacrolimus/Everolimus vs. Tacrolimus/MMF in Pediatric Heart Transplant Recipients Using the MATE Score
Acronym: TEAMMATE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Stanford University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kevin Daly, Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P00025970; PR160574 (Other Grant/Funding Number: U.S. Department of Defense); IND 127980 (Other: Food and Drug Administration)
Record Dates: First submitted 2017-12-18; First posted 2017-12-29 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Pediatric Heart Transplantation; Immunosuppression; Chronic Kidney Diseases; Cardiac Allograft Vasculopathy; Heart Transplant Failure and Rejection; Post-transplant Lymphoproliferative Disorder; Heart Transplant Infection
Keywords: heart transplantation; children; everolimus; tacrolimus; mycophenolate mofetil; randomized clinical trial
MeSH Terms: conditions — Renal Insufficiency, Chronic; Rejection, Psychology | interventions — Everolimus; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Multicenter open-label randomized clinical trial with randomization within 4 strata, defined by donor-specific antibody status and center annual transplant volume. There are 2 parallel groups of equal sizes for randomization: everolimus/low-dose tacrolimus and tacrolimus/mycophenolate mofetil.
Who Masked: Outcomes Assessor
Masking Description: The Coronary Angiography Core Laboratory readers will be blinded to treatment assignment and time point (study visit). The Adjudication Committee members will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Everolimus/Low-Dose Tacrolimus (Experimental): Everolimus approximately 0.6 mg/m2/dose taken by mouth every 12 hours for 30 months. Everolimus dose will be adjusted to achieve a trough concentration of 3-8 ng/ml.
  Tacrolimus 0.0125 mg/kg/dose by mouth every 12 hours for 30 months. (Tacrolimus dose will be adjusted to achieve a trough concentration of 3-5 ng/ml until subjects are 1 year post-heart transplant. After 1 year post-heart transplant the tacrolimus dose will be adjusted to achieve a trough concentration of 2.5-4.5 ng/mL.)
  Interventions: Drug: Everolimus; Drug: Tacrolimus
- Tacrolimus/Mycophenolate Mofetil (Active Comparator): Tacrolimus 0.05 mg/kg/dose by mouth every 12 hours for 30 months. (Tacrolimus dose will be adjusted to achieve a trough concentration of 7-10 ng/ml until subjects are 1 year post-heart transplant. After 1 year post-heart transplant the tacrolimus dose will be adjusted to achieve a trough concentration of 5-8 ng/mL.)
  Mycophenolate mofetil 600 mg/m2/dose by mouth every 12 hours for 30 months.
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Everolimus — Everolimus tablet
  Other Names: Zortress
  Arms: Everolimus/Low-Dose Tacrolimus
Drug: Tacrolimus — Tacrolimus capsule or liquid suspension
  Other Names: Prograf
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil capsule or liquid suspension
  Other Names: Cellcept
  Arms: Tacrolimus/Mycophenolate Mofetil

SUMMARY:
The TEAMMATE Trial will enroll 210 pediatric heart transplant patients from 25 centers at 6 months post-transplant and follow each patient for 2.5 years. Half of the participants will receive everolimus and low-dose tacrolimus and the other half will receive tacrolimus and mycophenolate mofetil. The trial will determine which treatment is better at reducing the cumulative risk of coronary artery vasculopathy, chronic kidney disease and biopsy proven-acute cellular rejection without an increase in graft loss due to all causes (e.g. infection, PTLD, antibody mediated rejection).

DETAILED DESCRIPTION:
Median survival after pediatric heart transplantation (HT) is 15 years in the current era. This means that a substantial fraction of patients transplanted during childhood fail to survive to adulthood, or require heart re-transplantation, because of complications related to heart transplant. These complications include heart transplant rejection, infection, coronary artery disease, post-transplant lymphoproliferative disorder (PTLD; a form of lymphoma seen in transplant recipients), and kidney failure. Most complications stem not from the heart transplant itself, but from the drugs commonly used to suppress the immune system in order to prevent rejection. In the US, tacrolimus (TAC) and mycophenolate mofetil (MMF), have emerged over the past decade as the standard of care for pediatric heart transplant immunosuppression. While pediatric survival has improved significantly in the era of TAC and MMF, post-HT complications remain a major problem that limits median survival to 15 years. Recently, everolimus (EVL) has emerged as a potential alternative immunosuppressant that may prevent rejection, coronary artery disease and kidney failure more effectively than TAC/MMF when administered in combination with low-dose tacrolimus (LDTAC). Preliminary studies suggest that EVL, and its first-generation analog sirolimus, are well tolerated in children after HT, regardless of whether it is started in response to coronary artery disease, in response to chronic kidney disease, or empirically 4-6 months after transplant in an effort to prevent the development of these complications1. However, studies are generally limited to single-center experiences using historical controls and have inadequate statistical power to demonstrate treatment differences. This will be the first multicenter randomized clinical trial of maintenance immunosuppression in pediatric heart transplantation to systematically evaluate the safety and efficacy of EVL with LDTAC vs. TAC/MMF to prevent long-term complications which lead to death/graft loss. The major adverse transplant event (MATE) score will serve as the primary endpoint to power the trial. Because no Food & Drug Administration (FDA)-approved immunosuppressants currently exist for children after heart transplant (all prescriptions are off-label) and market incentives to support a trial are limited, the investigators have funded the trial through a Fiscal Year 2016 Peer Reviewed Medical Research Program Clinical Trial Award sponsored by the Department of Defense office of the Congressionally Directed Medical Research Programs. It is worth noting that in contrast to adults, children have a substantially longer potential life expectancy if post-transplant complications can be minimized, making the prevention of late complications an urgent priority for the pediatric heart transplant community.

ELIGIBILITY:
Inclusion Criteria:

1. Orthotopic heart transplantation
2. Age < 21 years at time of transplant
3. Stable immunosuppression at the time of randomization with no contraindication to everolimus, tacrolimus, or mycophenolate mofetil
4. Planned follow-up at a study site for the 30 month duration of the study.
5. Subject or legal adult representative capable of providing informed consent (in general, assent will be sought for children aged 12 years or older).

Exclusion Criteria:

1. Multi-organ transplant (e.g. heart-lung or heart-liver).
2. Known hypersensitivity to everolimus, sirolimus, tacrolimus or mycophenolate mofetil (MMF), or to components of the drug products.
3. Patients on maintenance corticosteroid therapy exceeding a dose equivalent of prednisone 0.1 mg/kg/day at randomization.
4. High-risk for rejection defined as active rejection, recurrent (≥ 2 episodes of grade 2R rejection) cellular rejection, recurrent rejection (≥ 2 episodes of any grade) with hemodynamic compromise, steroid-resistant rejection or unresolved antibody-mediated rejection during the first 6 months post-heart transplant
5. Graft dysfunction (LVEF <40% or wedge pressure >22 mmHg or cardiac index <2.2 L/min/m2)
6. Stage 4 or 5 CKD (eGFR <30 ml/min/1.73 m2)
7. Moderate or severe proteinuria
8. Active infection requiring hospitalization or treatment dose medical therapy.
9. Patients with ongoing wound healing problems, clinically significant wound infection requiring continued therapy or other severe surgical complication in the opinion of the Site Principal Investigator.
10. Fasting Serum Cholesterol ≥300 mg/dL OR greater than or equal to 7.75 mmol/L, AND fasting triglycerides ≥2.5x the upper limit of normal (ULN). Note: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication, and reduction of serum cholesterol and triglyceride levels to below exclusion ranges is confirmed.
11. Uncontrolled diabetes mellitus.
12. Diagnosis of post-transplant lymphoproliferative disorder (PTLD) during the first 6 months post-heart transplant.
13. History of non-adherence to medical regimens.
14. Patients who are treated with drugs that are strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4) and cannot discontinue the treatment
15. Patients who are pregnant or breast-feeding or intend to get pregnant during the study period.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 211 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
EFFICACY: MATE-3 Score | 30 months post-randomization
  MATE-3 is a validated score ranging from 0 to 12. The score represents the cumulative burden of three major adverse transplant events: Coronary Artery Vasculopathy (CAV), Chronic Kidney Disease (CKD), and Biopsy-proven Acute Cellular Rejection (ACR)
SAFETY: MATE-6 Score | 30 months post-randomization
  MATE-6 is a validated score ranging from 0 to 24. The score represents the cumulative burden of all six major adverse transplant events: Coronary Artery Vasculopathy (CAV), Chronic Kidney Disease (CKD), Biopsy-proven Acute Cellular Rejection (ACR), pathologic diagnosis of Antibody-Mediated Rejection (AMR), Infection, and Post-Transplant Lymphoproliferative Disorder (PTLD)

SECONDARY OUTCOMES:
Efficacy: Overall patient survival | Up to 30 months post-randomization
  Freedom from death from any cause
Efficacy: Overall allograft survival | Up to 30 months post-randomization
  Freedom from death and re-transplantation
Efficacy: Change in kidney function | 0 to 6 months, 0 to 12 months, 0 to 30 months post-randomization
  Change in estimated glomerular filtration rate (eGFR) using the modified Schwartz equation
Efficacy: Freedom from CKD event | Follow-up through 30 months post-randomization
  Chronic Kidney Disease (CKD)
Efficacy: Freedom from CAV event | Follow-up through 30 months post-randomization
  Coronary Artery Vasculopathy (CAV)
Efficacy: Freedom from BP-ACR event | Follow-up through 30 months post-randomization
  Biopsy-proven Acute Cellular Rejection (ACR)
Efficacy: Freedom from composite failure | Follow-up through 30 months post-randomization
  The qualifying event is the earliest occurrence of death, graft loss, 2R/3R ACR rejection or rejection with HD
Efficacy: Lansky and Karnofsky scores | 18 and 30 months post-randomization
  Validated functional performance score, assigned by clinician assessment: Lansky score if < 16 years at randomization; Karnofsky if >=16 years at randomization
Efficacy: EuroQOL EQ-5D Y (Youth Version) | 18 and 30 months post-randomization
  Completed by study participant except for: EQ-5D-Y Proxy version will be used for children ≥ 4 years but less than 8 years at randomization or children ≥ 8 years who are unable to complete the EQ-5D-Y.
Safety: Freedom from AMR | Follow-up through 30 months post-randomization
  Pathologic diagnosis of Antibody-Mediated Rejection (AMR)
Safety: Freedom from infection | Follow-up through 30 months post-randomization
  Infection
Safety: Freedom from PTLD | Follow-up through 30 months post-randomization
  Post-Transplant Lymphoproliferative Disorder (PTLD)
Safety: Frequency and incidence of adverse events including, but not limited to, hyperlipidemia, anemia, thrombocytopenia, interstitial lung disease, aphthous stomatitis, proteinuria, and rash | Follow up through 30 months post-randomization
  These AEs will be reported as individual endpoints as well as a composite.
Safety: Freedom from Major Transplant Events (Composite) | Follow-up through 30 months post-randomization
  The qualifying event is the earliest occurrence of CKD, CAV, ACR, AMR, infection, and PTLD
Safety: Freedom from Level 2 severity CKD Event | Follow-up through 30 months post-randomization
  Chronic Kidney Disease
Safety: Freedom from Level 2 severity CAV Event | Follow-up through 30 months post-randomization
  Coronary artery vasculopathy
Safety: Freedom from Level 2 severity ACR Event | Follow-up through 30 months post-randomization
  Biopsy-proven Acute Cellular Rejection
Safety: Freedom from Level 2 severity AMR Event | Follow-up through 30 months post-randomization
  Pathologic diagnosis of Antibody-Mediated Rejection
Safety: Freedom from Level 2 severity Infection Event | Follow-up through 30 months post-randomization
  Infection
Safety: Freedom from Level 2 severity PTLD Event | Follow-up through 30 months post-randomization
  Post-transplant Lymphoproliferative Disorder
Efficacy: Freedom from composite of CAV, CKD, BP-ACR, or any CMV infection | Follow-up through 30 months post-randomization
  The event is the earliest occurrence of CAV, MATE CKD, BP-ACR, or any CMV infection.
Efficacy: Change in CKD stage | Baseline visit through 30 months post-randomization
  Change in chronic kidney disease stage where improvements in CKD stage can take on a negative value.
Efficacy: MATE-3 score where CKD score is calculated by change from baseline visit | Baseline visit through 30 months post-randomization
  MATE-3 score where the CKD score is the change in MATE-CKD score from baseline visit through 30 months post-randomization.
Efficacy: MATE-3 score where CKD score is replaced by change in CKD stage | Baseline visit through 30 months post-randomization
  MATE-3 score where the CKD score is replaced by change in CKD stage from baseline visit through 30 months post-randomization.
Efficacy: Composite score consisting of MATE CAV, MATE BP-ACR, change in MATE CKD score, and any CMV infection. | Baseline visit through 30 months post-randomization
  Efficacy: Composite score consisting of MATE CAV, MATE BP-ACR, change in MATE CKD score from baseline visit, and any CMV infection.
Efficacy: Composite score consisting of MATE CAV, MATE BP-ACR, change in CKD stage, and any CMV infection. | Baseline visit through 30 months post-randomization
  Efficacy: Composite score consisting of MATE CAV, MATE BP-ACR, change in CKD stage from baseline visit, and any CMV infection.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S Almond, MD, MPH, Study Chair — Stanford University; Kevin P Daly, MD, Study Chair — Boston Children's Hospital; Lynn A Sleeper, ScD, Principal Investigator — Boston Children's Hospital
Locations (25):
- United States (25):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Loma Linda University, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Congenital Heart Center, Gainesville, Florida
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Children's Healthcare of Atlanta Emory, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - Children's Hospital of New York, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Children's Health Dallas University of Texas Southwestern, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almond CS, Hoen H, Rossano JW, Castleberry C, Auerbach SR, Yang L, Lal AK, Everitt MD, Fenton M, Hollander SA, Pahl E, Pruitt E, Rosenthal DN, McElhinney DB, Daly KP, Desai M; Pediatric Heart Transplant Study (PHTS) Group Registry. Development and validation of a major adverse transplant event (MATE) score to predict late graft loss in pediatric heart transplantation. J Heart Lung Transplant. 2018 Apr;37(4):441-450. doi: 10.1016/j.healun.2017.03.013. Epub 2017 Mar 24. PMID 28465118
- [Background] Castleberry C, Ziniel S, Almond C, Auerbach S, Hollander SA, Lal AK, Fenton M, Pahl E, Rossano JW, Everitt MD, Daly KP. Clinical practice patterns are relatively uniform between pediatric heart transplant centers: A survey-based assessment. Pediatr Transplant. 2017 Aug;21(5). doi: 10.1111/petr.13013. Epub 2017 Jul 3. PMID 28670871
- [Background] Almond CS, Sleeper LA, Rossano JW, Bock MJ, Pahl E, Auerbach S, Lal A, Hollander SA, Miyamoto SD, Castleberry C, Lee J, Barkoff LM, Gonzales S, Klein G, Daly KP. The teammate trial: Study design and rationale tacrolimus and everolimus against tacrolimus and MMF in pediatric heart transplantation using the major adverse transplant event (MATE) score. Am Heart J. 2023 Jun;260:100-112. doi: 10.1016/j.ahj.2023.02.002. Epub 2023 Feb 23. PMID 36828201
- [Derived] Almond CS, Daly KP, Albers EL, Alejos JC, Ameduri R, Auerbach SR, Barkoff L, Barnes AP, Bock MJ, Butto A, Carlo WF, Castleberry CD, Chrisant MR, Deshpande SR, Dreyer WJ, Everitt MD, Feingold B, Gonzales S, Hollander SA, Kindel SJ, Klein GL, Lal AK, Lamour JM, Lee J, Lu M, Lytrivi ID, Miyamoto SD, Pahl E, Peng DM, Ryan TD, Singh TP, Su JA, Sutcliffe DL, Ybarra AM, Zangwill S, Rossano JW, Sleeper LA; TEAMMATE Trial Investigators. Everolimus and Low-Dose Tacrolimus After Heart Transplant in Children: A Randomized Clinical Trial. JAMA. 2025 Oct 21;334(15):1339-1348. doi: 10.1001/jama.2025.14338. PMID 40960806
- [Derived] Grimm K, Lehner A, Fernandez Rodriguez S, Orban M, Fischer M, Rosenthal LL, Jakob A, Haas NA, Dalla Pozza R, Kozlik-Feldmann R, Ulrich SM. Conversion to everolimus in pediatric heart transplant recipients is a safe treatment option with an impact on cardiac allograft vasculopathy and renal function. Clin Transplant. 2021 Mar;35(3):e14191. doi: 10.1111/ctr.14191. Epub 2020 Dec 30. PMID 33315277